CLINICAL TRIAL: NCT02272283
Title: Optical Coherence Tomography Guided Percutaneous Coronary Intervention With Nobori Stent Implantation in Patients With Non ST Segment Elevation Myocardial Infarction
Brief Title: Optical Coherence Tomography Guided Percutaneous Coronary Intervention With Stent Implantation
Acronym: OCTACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Lisbeth Antonsen, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20110030
Record Dates: First submitted 2014-10-15; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: PCI optimization; Coronary Remodeling; Drug-Eluting Stent; Optical Coherence Tomography; Intravascular Ultrasound; Strut Coverage; Strut Apposition; Vascular Healing Pattern
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angio-guided PCI (Active Comparator): Patients allocated to "angio-guided PCI" are having Percutaneous Coronary Intervention (PCI) with stent implantation guided by routine angiography alone.
  Documentary (comparator) intravascular imaging with Optical Coherence Tomography (OCT) and Intravascular Ultrasound (IVUS) is performed. The PCI-operator is blinded to the image aquisitions, and the analysis is performed offline later.
  Interventions: Device: Percutaneous coronary intervention with Nobori biolimus-eluting stent implantation
- OCT-guided PCI (Experimental): After obtaining an angiographic optimal result, patients allocated to "OCT-guided PCI" have guiding Optical Coherence Tomography (OCT) and Intravascular Ultrasound (IVUS) performed. Online image interpretation is performed by a dedicated OCT-analyst and the PCI-operator. If the OCT reveals; 1) under expansion of the stent with a minimal stent area (MSA) <90% of the distal/proximal reference vessel lumen area and/or; 2) significant acute incomplete stent apposition (defined as more than or equal to 3 stent struts detached >140 microns from the underlying vessel wall), and/or; 3) edge dissection(s) causing significant reduction in minimal lumen area(s) (MLA <4 mm2) and/or, 4) significant residual stenosis (MLA <4 mm2) at the proximal and/or distal reference segment(s), additional intervention is encouraged. The degree of optimization based upon OCT findings is left to the judgement of the PCI-operator.
  Interventions: Device: Percutaneous coronary intervention with Nobori biolimus-eluting stent implantation

INTERVENTIONS:
Device: Percutaneous coronary intervention with Nobori biolimus-eluting stent implantation — The third-generation biodegradable polymer Nobori biolimus-eluting stent is implanted in all patients

SUMMARY:
Coronary artery disease is one of the most prevalent diseases in the western countries.

A waxy substance called plaque can build up inside the coronary arteries. Over time, plaque can harden or rupture, and cause narrowing (stenosis) of the arteries and reduce the flow of oxygen-rich blood to the heart.

The standard treatment of symptomatic coronary stenosis is percutaneous coronary intervention (PCI) with balloon dilation followed by stent implantation.

A stent is a small metallic grid that stabilizes the coronary vessel wall after the balloon dilation.

Currently, drug-eluting stents (DES) are the most widely used stent types. DESs consist of a metallic backbone and an antiprolifetive drug-coating bound by a polymer (glue). These devices have reduced the incidence of excessive formation of new tissue (in-stent restenosis) dramatically in comparison with previously used bare-metal stents.

However, there are "safety concerns" with DES, since later thrombotic events have been reported.

On one hand excessive tissue formation inside the stent can cause in-stent restenosis, and on the other hand insufficient coverage of the stent can cause persistently exposed metalllic material that can induce platelet aggregation and thrombus-formation.

The etiology to stent thrombosis is multifactorial. Possible predisposing factors are, among others: 1) hypersensitivity towards the polymer-coating, which may induce delayed healing inside and around the stent, and 2) insufficient contact between the stent and the underlying coronary vessel wall (incomplete stent apposition), which may cause flow-disturbance and delayed healing.

Delayed healing causes persistently exposed metallic material that can induce platelet aggregation and thrombus-formation.

The Nobori stent is a new-generation DES, coated with a thin layer of drug and a bioabsorbable polymer. The drug is localized on the outer side of the stent, and decreases the release of drug to the blood circulation. The bioabsorbable polymer is degraded after 6-9 months after implantation, and decreases the risk of hypersensitivity-reactions in the vessel wall.

The improved pharmacokinetic profile of the stent is thought to improve the healing pattern.

At routine coronary angiography, a small plastic tube is inserted in the femoral artery under local anesthesia. Thin, flexible catheters are then advanced through the artery system (femoral artery and aorta) to the coronary arteries. Contrast is injected in to the blood stream by the catheters, and the arteries are depicted by a special X-ray technique during dye-release. By angiography, the outer sides of the coronary arteries are visualized, and balloon dilations and stent implantations are guided by this standard technique.

Newer studies have documented that stent placement and expansion is superiorly visualized if supplementary intravascular imaging is performed during stent implantation.

Small imaging catheters are wired through the vessel after stent implantation, and film the stent retrogradely through the vessel.

Intravascular ultrasound (IVUS) visualizes the complete vessel wall by use of sound waves, and stent expansion is evaluated in detail.

Optical coherence tomography (OCT) is a newer light-based, high-resolution technology. The technique can depict every thread (strut) from the stent, enabling visualization of both contact between struts and underlying vessel wall immediately after the procedure, and strut coverage at follow-up.

The purpose of this study is to determine whether OCT-guided PCI can improve healing and coverage of the stent in comparison with routine angiographic guidance alone in patients indicating PCI due to myocardial infarction.

If OCT-guidance improves coverage of the stent, this might lower the later thrombotic risk.

Patients hospitalized due to myocardial infarction are randomized either to OCT-guided or angio-guided stent implantation in the present study. In both groups the Nobori stent is implanted according to standard techniques. In the angio-guided group, implantations are guided by angiography alone. OCT- and IVUS analysis are performed after an angiographic optimal result for documentary reasons. The operator is blinded towards the image findings, and analysis is performed offline later.

In the OCT-guided group, both OCT and IVUS analysis is interpreted immediately after the acquisition. If stent apposition and/or expansion is deemed suboptimal, additional balloon dilation and/or stenting is performed. In case of OCT-driven stent optimization, a documentary OCT and IVUS is performed to document the final result.

Patients are readmitted 6 months later for a control angiogram inclusive OCT to assess stent coverage.

Furthermore, patients are readmitted 12 months after the index procedure for a control angiogram including OCT and IVUS to assess dynamic vessel wall responses.

DETAILED DESCRIPTION:
Drug-eluting stents (DES) have reduced the rate of in-stent restenosis dramatically in comparison with bare-metal stents (BMS). Still, there are "safety concerns" in form of late and very late stent thrombosis.

Multifactorial predictors may be associated with later thrombotic events, but delayed arterial healing has been documented the most powerful predisposing factor in previous histo-pathological studies. Culprit lesions in patients having DES-implantation due to myocardial infarction are associated with substantial delay in arterial healing in comparison with patients having DES-implantation due to stable coronary artery disease.

Numerous procedural factors are also of significant importance with regard to sufficient coronary vessel wall healing. Particularly, acute incomplete stent apposition (ISA) is a strong procedural risk factor for delayed coverage.

Optical coherence tomography (OCT) is a high-resolution intravascular imaging modality, which enables detailed in-vivo assessment of the immediate stenting result and the vascular healing pattern, including strut coverage, at follow-up.

Some procedural factors can be modified using OCT-guidance, potentially leading to a decrease in the proportion of uncovered struts at follow-up.

The hypothesis of the study is that OCT-guided PCI can reduce the incidence of acute and late ISA, and thereby provide improved strut coverage following Nobori-stent implantation.

The objective of this study is to assess whether OCT-guided optimization following Nobori stent implantation in patients with Non ST segment Elevation Myocardial Infarction (NSTEMI) improves the coronary vascular response in comparison with routine angiographic guidance alone.

The present study is designed as a prospective, randomized trial conducted at a single center (Odense University Hospital). One-hundred patients were enrolled (Between August 2011 and May 2013). Prior to the PCI procedure, patients were loaded with a 300 mg dose of aspirin, and a loading dose of 180 mg ticagrelor. An unfractionated heparin dose (70 IU/kg) was administered just before the PCI-procedure. In all cases the third-generation biolimus-eluting stent (Nobori, Terumo, Tokyo, Japan) was implanted.

Stents were implanted according to standard techniques. Recommended post-procedure dual antiplatelet regimens were 75 mg aspirin daily lifelong and 90 mg ticagrelor twice daily for 1 year.

Post-implantation, after acquisition of an angiographic optimal result, patients were randomly assigned 1:1 to either: 1) OCT-guided PCI, or 2) angio-guided PCI. Random assignments were distributed in sealed envelopes.

Both treatment arms had post-procedure OCT and IVUS performed after administration of 200 micrograms of intracoronary nitroglycerin. It was not possible to blind the operator, investigator or patient for the allocated implantation technique, but the operator was blinded to the post-procedure OCT- and IVUS images in the angio-guided group, as the operator screen-side was turned off, and the entire pullbacks remained uncommented on. In the OCT-guided group, images were interpreted online by a dedicated OCT-analyst and the PCI-operator.

If the post-procedure OCT revealed: 1) under expansion of the stent with a minimal stent area (MSA) <90% of the distal/proximal reference vessel lumen area, and/or 2) significant acute ISA (defined as more or equal to 3 struts per cross sectional area detached more than 140 microns (thickness of strut + drug/polymer coating)) from the underlying vessel wall, and/or 3) edge dissection(s) causing significant reduction in minimal lumen area(s) (MLA<4 mm2) and/or 4) significant residual stenosis (MLA<4 mm2) at the proximal and/or distal reference segment(s) additional intervention was encouraged. The degree of optimization based upon OCT findings was left to the judgement of the PCI-operator.

Patients were scheduled for both a 6-months clinical and invasive (including angiogram and OCT) and a 12-months clinical and invasive (including angiogram, OCT and IVUS) follow-up.

Prior to follow-up imaging, 5,000 IU of unfractionated heparin and 200 micrograms of intracoronary nitroglycerin was administered.

OCT was performed both post-procedure, at 6-months and at 12-months using a frequency-domain OCT system (C7-XR or Ilumien system). A 2.7 Fr C7 Dragonfly imaging catheter flushed with 20 ml undiluted contrast was used.

Motorized pullback was performed at a pullback rate of 20 mm/s throughout the stent.

Quantitative OCT analysis is performed using the LightLab OCT proprietary software (Offline Review Workstation). Analysis is performed by one dedicated OCT-analyst, who is blinded to the implantation technique, when assessing 6-months images for strut coverage.

An inter-observer reliability analysis of apposition and coverage will be provided.

Lesions are analyzed at the cross sectional level with an interval of 1 mm (every 5 frames).

Struts devoid of coverage at any part are deemed "uncovered". The neointimal thickness is measured for all covered struts (the thickness is measured as the distance between the endoluminal side of the strut from the midpoint of its long axis and the intersection of the lumen contour with a straight line between the endoluminal side of the strut and the gravitional center of the vessel). Apposition is assessed by measuring the distance between the center of the endoluminal strut side and the gravitional center of the vessel (malapposed strut = detached more than 140 microns from the underlying vessel wall).

Malapposition distances and areas are also traced. The percentage of malapposed and/or uncovered struts are calculated as the number of malapposed and/or uncovered struts/total number of struts in all cross sections of the lesion, multiplied by 100.

The IVUS system (Boston Scientific) utilized a 40 MHz, 2.6 Fr IVUS catheter (Atlantis SR Pro). Image acquisition using automated transducer pullback at 0.5 mm/s was performed from at least 10 mm distal to 10 mm proximal of the stented segment.

Offline analysis is performed with a computerized planimetry program (EchoPlaque). For each 1 mm of axial length, lumen and external elastic membrane (EEM) areas are traced. Stent and reference site parameters (areas and volumes) are calculated. Remodeling (based on baseline and 12-months analysis) is assessed.

SPSS version 22.0 (SPSS Inc., Chicago Illinois) is used for the statistical analysis. All tests are two-tailed, and a p-value <0.05 is considered statistically significant. Categorical data will be presented as numbers and frequencies, and compared with chi-square or Fisher´s exact statistics. Continuous data will be presented as mean +- SD and compared with the Student´s t-test. If the distributions are skewed, a non-parametric test will be performed, and the median with an interquartile range will be provided.

The primary and secondary endpoints will be assessed by the Kruskal-Wallis test, and an ordered logistic regression analysis adjusted for confounders will be provided.

Powercalculation: A powercalculation with an expected frequency of 0.66 and 0.90 covered struts after 6 months in the angio-guided and OCT-guided group, respectively, shows that 43 patients are to be included in each arm to reach statistical significance. With 43 patients in each treatment arm and a two-sided statistical significance level of 0.05, the study will have a power of 0.8 to show a proportion of 0.66 and 0.90 covered struts at 6-months follow-up in the angio- and OCT-guided group, respectively. With an expected dropout of 14% due to invasive non-compliance and with subject to suboptimal imaging quality, 100 patients are to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* A Non ST segment Elevation Myocardial Infarction (NSTEMI) had been diagnosed
* A de novo lesion (more than or equal to 50% dimater stenosis) had been visualized on coronary angiography
* A Percutaneous Coronary Intervention with Drug-Eluting Stent (DES) implantation was indicated

Exclusion Criteria:

* Patients included in other randomized trials
* Lifeexpectancy <1 year
* Allergy to aspirin, clopidogrel, ticagrelor and prasugrel
* Allergy to limus-agents
* Ostial lesions (not possible to flush by OCT)
* S-creatinin >170 micrograms/l
* Tortuous and extremely calcified lesions where intravascular imaging is deemed associated with an increased risk for the patient
* Very long lesions (due to the limited pullback length of the OCT system)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Proportion of uncovered struts | At 6-months follow-up OCT
  For each patient/stented segment: Number of uncovered struts divided by the total number of struts, multiplied by 100

SECONDARY OUTCOMES:
Number/Incidence of OCT-detected edge dissections | Assessed immediately after the stent implantation
  The frequency of angiographically silent edge dissections will be described
Spontaneous healing course of OCT-detected edge dissections | At 6-months follow-up OCT
  The number of residual dissection flaps and/or vessel wall disruptions will be described in relation to findings of edge dissections immediately after stent implantation
Dynamic coronary evaginations | At 6- and 12-months OCT
  Coronary evaginations are outward bulges of the vessel wall between struts. For each evagination observed, a "depth" and an "area" will be measured. Number and magnitude of coronary evaginations will be measured for each patient. Frequencies and magnitudes of these features at 6-months will be compared with frequencies and magnitudes of these features at 12-months
Peri-stent coronary vessel wall remodeling | IVUS immediately after stent implantation and after 12-months
  Remodeling will be assessed using IVUS, by measuring the serial changes in external elastic membrane cross sectional area between these 2 time points

REFERENCES:
- [Derived] Antonsen L, Thayssen P, Maehara A, Hansen HS, Junker A, Veien KT, Hansen KN, Hougaard M, Mintz GS, Jensen LO. Optical Coherence Tomography Guided Percutaneous Coronary Intervention With Nobori Stent Implantation in Patients With Non-ST-Segment-Elevation Myocardial Infarction (OCTACS) Trial: Difference in Strut Coverage and Dynamic Malapposition Patterns at 6 Months. Circ Cardiovasc Interv. 2015 Aug;8(8):e002446. doi: 10.1161/CIRCINTERVENTIONS.114.002446. PMID 26253735